

## Patient consent form - clinical trial

| ш | ie: Study of advance care planning will | n older pallents | s who have rehal la | liure |
|---|---|---|---|---|
| Na | me of Researcher: Dr Peter O'Hallora | ın | | |
| Centre Number (please circle): | | | | |
| Participant Identification Number for this trial: | | | | Please<br>initial<br>box |
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had my questions fully answered. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my health care being affected. | | | |
| 3. | I understand that relevant members of the research team will look at my medical records to collect information on my medical condition and also about my use of health services over the twelve months of the research. I give permission for these individuals to have access to my records. | | | |
| 4. | | | | the |
| 5. | I agree to take part in the above study. | | | |
| | Name of Participant (CARS) | Doto | Ciana | aturo |
| | Name of Participant (CAPS) | Date | Signa | ature |
| Name of person taking consent (CAPS) | | Date | <br> Signa | Signature |